CLINICAL TRIAL: NCT04979871
Title: Kinetics and Stability of Anti-SARS-CoV-2 Antibodies and Virus Neutralization After COVID-19 Vaccination in a Swiss Cohort
Brief Title: SARS-CoV-2 Antibodies and Virus Neutralisation in a Cohort Vaccinted Against COVID-19
Acronym: DER-CoV2-001
Status: Completed | Type: Observational
Sponsor: University of Zurich (Other)
Responsible Party: Principal Investigator, Pal Johansen, Professor Dr. sc., University of Zurich
Other Study IDs: DER-CoV2-001; BASEC Nr (Other: 2021-01361)
Record Dates: First submitted 2021-07-25; First posted 2021-07-28 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2023-05

CONDITIONS: Vaccine Reaction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Biospecimen Retention: Samples Without DNA — Serum
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Venous bleeding — Blood samples collected 5 times with approx. 2-4 weeks interval

SUMMARY:
Analysis of SARS-CoV-2 antibodies and serum virus neutralisation in vaccinated heath care personnel. Analysis of virus neutralisation as a function of age, gender, and history of COVID-19 infection.

DETAILED DESCRIPTION:
This study is an observational study with subsequent use of coded biological material. Sera of Universitiy Hospital of Zurich (USZ) personnel vaccinated with BNT162b2 (BioNTech/Pfizer) was analyzed for SARS-CoV-2 specific antibodies and virus neutralization.

Serum was analysed for virus-specific IgG and IgA using ELISA kits from Euroimmun (Kriens, Switzerland) according to the manufacturer's instruction. IgG was determined with the quantitative Anti-SARS-CoV-2 Quantivac kit and IgA was determined with the semi-quantitative Anti-SARS-CoV-2 kit The kits determine antibodies against the spike-1 protein. The sera were not diluted and not heat-inactivated prior to testing. The developed 96-well plates were analysed by reading absorbance at 450 nm using an ELx808 ELISA reader from BioTek Instr. Inc.

In addition, a SARS-CoV-2 neutralization assay was developed at the department. In this Tissue Culture Infection Dose (TCID) assay, Vero cells were infected with live SARS-CoV-2, and sera were added at various dilutions to test the potential to neutralize viral infection. The assay was conducted in a biosafety level 3 lab. Briefly, VERO-E6 cells were grown overnight to ca. 80-90% adherence in flat-bottom 96-well cell culture plates. The SARS-CoV-2 was then mixed in round-bottom 96 well titre plates with 2-fold serial dilutions of serum and incubated. The virus-serum mixture was then added to the VERO-E6 cell, and the cultures were incubated again. After three days, the cultures were fixed by addition of paraformaldehyde and stained with crystal violet for visualisation of cytotoxicity. The highest serum dilution preventing infections of the cells was defined as the neutralization titre.

ELIGIBILITY:
Inclusion Criteria:

* Employed at the USZ Department of Dermatology
* Vaccinated against Covid-19 at USZ
* Male and female persons of any age
* Serum samples collected in 2020 or until June 11th 2021
* The subject was informed and gave his/her consent to the research project (non-coded samples and data) and to publish data obtained from analysis of own biological samples

Exclusion Criteria:

* Known clinical relevant disease, e.g. immune suppressed by drugs or disease
* Documented objection of subsequent use and publication of biological samples and personal health data

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Approximately 250 blood samples from 50 vaccinated persons working in the USZ Department of Dermatology were collected in 2020 and 2021. All individuals recieveid either one or two doses of BNT162b2 (BioNTech/Pfizer) vaccine between January 2021 and June 2021. The persons providing blood samples (study subjects) were recruited by a general email (in English) to all members of the research unit of the Department of Dermatology (cf. Appendix). The sera were frozen and kept at the Dermatology biobank. The samples are labelled with subjects initials and date of sampling.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2021-07-22 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Immunity to Covid-19 vaccines | July 2021 through September 2021
  Analysis SARS-CoV-2 immunity with ELISA anti-S1 IgG and IgA assay and tissue-culture infection dose (TCID) neutralisation assays

CONTACTS AND LOCATIONS:
Overall Officials: Pål Johansen, Prof, Principal Investigator — University of Zurich, Dept. Dermatology
Locations (1):
- Univeristy Hospital Zurich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No
Study protocol is shared

REFERENCES:
- [Derived] Sosic L, Paolucci M, Duda A, Hasler F, Walton SM, Kundig TM, Johansen P. Kinetics and persistence of anti-SARS-CoV-2 neutralisation and antibodies after BNT162b2 vaccination in a Swiss cohort. Immun Inflamm Dis. 2022 Mar;10(3):e583. doi: 10.1002/iid3.583. Epub 2021 Dec 29. PMID 34965032